CLINICAL TRIAL: NCT04561986
Title: A Randomized Controlled Open-label Multi-center Study to Assess the Efficacy of TCZ in Treatment of Late/Chronic Active Antibody-mediated Rejection in Kidney Transplant Recipients
Brief Title: TocIlizumab in Late/Chronic Active Antibody-mediated Rejection in Kidney Transplant Recipients
Acronym: INTERCEPT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Karolinska University Hospital (Other); Uppsala University Hospital (Other); Skane University Hospital (Other); The Swedish Research Council (Other Government); Hospital del Mar (Other); Hospital Universitario Doctor Peset (Other); Complexo Hospitalario Universitario de A Coruña (Other); Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Seema Baid-Agrawal, Associate Professor and Consultant Nephrologist, Transplantation Center, Sahlgrenska University Hospital, Gothenburg, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-004302-10; 2024-510615-29-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-03; First posted 2020-09-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Antibody-mediated Rejection
Keywords: Kidney transplant; Chronic rejection; Antibody-mediated rejection; Graft function; Donor specific antibodies (DSA); Transplant-specific well-being; Adherence
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Standard of care (SOC) + tocilizumab (TCZ) (Active Comparator): SOC, as below + TCZ (162 mg every week, subcuataneous administration)
  Interventions: Drug: Tocilizumab
- Arm B: SOC (No Intervention): Tacrolimus (target concentration 6 ±1 µg/L) + MPA (1.5-2 g/day as tolerated) + prednisolone (not less than 5 mg/day), all oral administration

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab is a recombinant humanized monoclonal antibody directed against the human interleukin-6 (IL-6) receptor
  Other Names: RoActemra
  Arms: Arm A: Standard of care (SOC) + tocilizumab (TCZ)

SUMMARY:
This multi-center study is an investigator-driven randomized controlled parallel group open-label clinical trial designed to evaluate the efficacy of addition of anti-IL-6 antibody tocilizumab (TCZ) to the standard of care (SOC) treatment as compared to the SOC alone in reducing the decline of graft function in kidney transplant recipients with late or chronic antibody-mediated rejection (AMR). A total of 50 recipients will be allocated to receive either TCZ (n=25) added to the standard of care (SOC) or SOC alone (n=25) for a period of 24 months. Patients will be followed for an additional 12 months. Protocol kidney graft biopsies will be performed at 12 and 24 months. The primary outcome is the mean rate of change in graft function as assessed by estimated glomerular filtration rate (eGFR) slope from baseline to 24 months after start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has given their written informed consent to participate in the study
2. Recipient of living donor or deceased donor kidney transplant
3. Age ≥18 years
4. At least 6 months post-transplantation at randomization
5. Biopsy-proven diagnosis of late active or chronic active ABMR (≥ 6 months after transplantation) according to the Banff 2022 criteria in index biopsy
6. eGFR ≥20 ml/min/1.73 m2
7. Epstein-Barr Virus (EBV) IgG-positive
8. For female participants of childbearing potential:

   * use of adequate contraception and a negative pregnancy test
9. Subject known to have COVID-19 previously must meet all of the following conditions:

   * Asymptomatic for at least 1 month before the start of screening
   * Re-established on background immunosuppressants for at least 1 month prior to the randomization

Exclusion Criteria:

1. Recipient of multi-organ transplants
2. De novo or recurrent renal disease that is considered to be the predominant cause of the current graft dysfunction
3. Active viral infections such as BK virus (BKV), cytomegalovirus (CMV), EBV, COVID-19, hepatitis C virus (HCV) or hepatitis B virus (HBV) infections based on polymerase chain reaction (PCR) testing
4. Ongoing serious infections as per Investigator's opinion
5. History of recurrent infections requiring hospitalization
6. Active tuberculosis (TB)
7. Latent untreatedTB (positive QuantiFERON-TB-Gold test, Chest X-ray)
8. Abnormal liver function tests alanine transaminase (ALT), aspartate transaminase (AST), bilirubin > 1.5 x upper limit of normal)
9. Other significant liver disease as per Investigator's opinion
10. Neutropenia (<2 x109/L) or thrombocytopenia (<100 x109/L)
11. Signs of post-transplant lymphoproliferative disorder
12. Signs of malignancy. Exceptions are basal cell carcinoma/squamous cell carcinoma or non-malignant melanoma
13. History of malignancy, unless subject has been considered to have fully recovered from malignancy since > 2 years, without any signs of relapse
14. History of diverticulitis, inflammatory bowel disease or gastrointestinal perforation
15. Ongoing alcohol or illicit substance abuse
16. Serious medical or psychiatric illness likely to interfere with participation in the study as per Investigator's opinion
17. Mental inability or reluctance that results in difficulties in understanding the meaning of study participation
18. Woman of childbearing potential who is unwilling/unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 8 weeks after the last dose of study drug
19. Woman with a positive pregnancy test or who is pregnant or breastfeeding
20. Current or recent (within last 3 months) participation in another clinical drug trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in eGFR at 24 months | Baseline and 24 months
  Comparison of eGFR decline (eGFR slope) from baseline at 24 months after start of treatment in the two arms. The eGFR will be assessed by measured creatinine values using MDRD formula in mL/min/1.73m^2. MDRD formula is based on age, sex, ethnicity, and serum creatinine (in mg/dl) and eGFR values are calculated as follows: GFR in mL/min per 1.73 m^2 = 175 x Serum Cr^1.154 x age^-0.203 x 1.212 (if patient is black) x 0.742 (if female).

SECONDARY OUTCOMES:
Composite risk prediction score iBox | baseline and upto 24 months
  Efficacy of the treatment regimen by assessing the iBox score
Incidence of adverse and serious events related to TCZ treatment | up to 25 months
  Assessments of incidence of any side effects including infectious complications associated with TCZ therapy
Change in Donor-specific anti-HLA antibodies (DSA) | baseline and up to 36 months
  Change in DSA from baseline based on luminex assessments every 12 months
Histologic changes in protocol biopsy | baseline and up to 24 months
  Histologic changes at 12 and 24 months will be compared with those in the baseline biopsies. If the criteria for active AMR are no longer fulfilled in the follow-up biopsies, response to therapy is assumed. The response will be assessed as a yes/no categorical variable. In all biopsies, which still meet the required criteria for active AMR, means of individual Banff lesion scores will be compared between the baseline biopsy and the 12- and 24-months biopsies
Changes in proteinuria | baseline and up to 36 months
  Assessed by urine albumin creatinine ratio (UACR) at baseline and every 12 months
Renal function assessed by measured GFR (mGFR) | baseline and up to 36 months
  Changes from baseline in renal function as assessed by mGFR using iohexol clearance
Renal function assessed by eGFR | baseline and up to 36 months
  Changes from baseline in renal function at 12 and 36 months after start of treatment, as assessed by eGFR (CKD-EPI)
Patient survival | up to 36 months
  Incidence of patient survival at 12, 24 and 36 months after start of treatment
Death-censored graft survival | up to 36 months
  Incidence of death-censored graft survival at 12, 24 and 36 months after start of treatment
Possible change in experienced transplant-specific well-being and symptom burden | upto 36 months
  Assessed using a validated self-reported questionnaires at baseline and every 12 months
Possible change in experienced perceived threat of the risk of graft rejection | upto 36 months
  Assessed using a validated self-reported questionnaires at baseline and every 12 months
Possible change in adherence to immunosuppressive medications | upto 36 months
  Assessed using a validated self-reported questionnaires at baseline and every 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Seema Baid-Agrawal, MD, FASN, Principal Investigator — Transplant Center, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (8):
- Spain (4):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Marqués de Valdecilla Research Institute, Santander
  - Hospital Universitario Dr. Peset, Valencia
- Sweden (4):
  - Skåne University Hospital, Malmo, Skåne County
  - Transplant Center, Sahlgrenska University Hospital, Gothenburg, Vastra Gotaland Regioin
  - Karolinksa University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Streichart L, Felldin M, Ekberg J, Mjornstedt L, Lindner P, Lennerling A, Brocker V, Molne J, Holgersson J, Daenen K, Wennberg L, Lorant T, Baid-Agrawal S. Tocilizumab in chronic active antibody-mediated rejection: rationale and protocol of an in-progress randomized controlled open-label multi-center trial (INTERCEPT study). Trials. 2024 Mar 22;25(1):213. doi: 10.1186/s13063-024-08020-0. PMID 38519988